CLINICAL TRIAL: NCT03290066
Title: Effectiveness of Kinesiotaping in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena Estebanez de Miguel, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UZaragoza
Record Dates: First submitted 2017-09-12; First posted 2017-09-21 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Kinesio Taping
MeSH Terms: interventions — Athletic Tape; Self Care

STUDY DESIGN:
Intervention Model Description: Each woman will be assigned to a sequence of treatments, including two treatments (kinesiotape and usual dysmenorrhea treatment). The sample will be randomized in two different sequences of treatments (kinesiotape/usual treatment or usual treatment/kinesiotape)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Active Comparator): Kinesiotape will be applied as a self-treatment. All participants will be instructed in an indvidual session and will receive a tutorial video to remember the kinesiotaping procedure. 3 band of a special and hypoallergenic tape (Kinematix Tex) will be attached to the abdominal (2 strips) and lower back (1 strip).
  Patients will be taped for four days , ıt will start at the beginning of the menstruation.
  Interventions: Device: kinesiotape
- Usual care (Active Comparator): Participants will use the usual self-care for primary dysmenorrhea. It will start at the beginning of the menstruation.
  They will note the treatment indicating the dosage in a calendar.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: kinesiotape — For the Kinesio taping group, a piece of Kinesio tape 5 cm in width and 7-8 cm in length will be applied right from below the navel and will reach to where the pubic hair begins, and another piece of tape 10 cm in length will be applied to make a cross shape with the first piece. A tape of 20cm in length will be placed horizontally to the lower back.
  Arms: Kinesiotape
Other: Usual care — Participants will note the usual self-care used to relief pain (NSAIDs, heat, massage therapy.....).
  Other Names: self-care
  Arms: Usual care

SUMMARY:
Determine the effectiveness of kinesiotaping on pain in primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as cramping pain in the lower abdomen occurring just before or during menstruation, in the absence of other diseases.

Dysmenorrhea is estimated to occur in 45% to 90% of women of reproductive age. It is a common cause of absenteeism and reduced quality of life in women.

Treatment for dysmenorrhoea aims to relieve pain or symptoms either by affecting the physiological mechanisms behind menstrual pain (such as prostaglandin production) or by relieving symptoms.

First line treatment for dysmenorrhoea is oral contraceptives, non-steroidal anti-inflammatory drugs, paracetamol or aspirin. However these present side effects and some women have contraindications to these treatments. Consequently, it´s necessary to study alternative treatments to drug treatments. Alternative treatments like heat, massage therapy, acupuncture also are used.

The Kinesiotaping uses an adhesive elastic cotton tape color invented by Dr. Kase in the 1970s. It is water resistant and retains its properties up to 5 days.

It has the characteristic to cause elevation of the epidermis and thereby reduce the pressure on the mechanoreceptors below the dermis. This would have the effect of reducing nociceptive stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting menstrual pain, 4 or more in VAS.
* Have attended gynecological examination in the past 18 months and had ever diagnosed as having a gynecological disorder different from primary dysmenorrhea
* Not have been diagnosed with secondary dysmenorrhea
* Regular menstrual cycles (cycle typical range of 21 to 35 days)
* Do not use an intrauterine contraceptive device (IUD) or taking oral contraceptive pills
* Nulliparous
* Ability to complete questionnaires in Spanish.

Exclusion Criteria:

* Women with mild dysmenorrhea (pain lower 4 in a numeric pain scale range 0-10);
* Women with irregular or infrequent menstrual cycles (outside the typical range of cycle 21 to 35 days);
* Women using an intrauterine contraceptive device (IUD) or taking oral contraceptive pills.
* Women who suffer from diseases diagnosed added
* Women to which it has undergone a surgical procedure for the treatment
* Provide skin lesions in the abdominal wall or in lumbar region
* Use or abuse of drugs or alcohol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in menstrual pain with Visual Analogic Scale (VAS) | Participants will be followed for 2 menstrual cycles, an expected average of 3 months. Evaluations will be performed before, and just after 2 hours, 8 hours, 12 hours, 24 hours, and 48 hours after treatment
  VAS is a method of representing subjects' pain on a 10 cm linear scale. In this study, a score of 0 means 'a very low degree of pain' and 10 means 'a very high degree of pain.'

SECONDARY OUTCOMES:
Patient satisfaction with Visual Analogic Scale (VAS) | Participants will be followed for 2 menstrual cycles. Evaluations will be performed at the end of each treatment, when menstrual pain disappears (4-5 days after the beginning of the menstrual bleeding).
  Participants will note the self-care applied to relief menstrual pain indicating the VAS is a method of representing subjects' satisfaction with treatment on a 10 cm linear scale. In this study, a score of 0 means 'a very low degree of satisfaction with treatment' and 10 means 'a very high degree of satisfaction with treatment.'

CONTACTS AND LOCATIONS:
Overall Officials: Elena Estebanez de Miguel, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Elena Estebanez de Miguel, Zaragoza, Spain